CLINICAL TRIAL: NCT06803147
Title: "Less-is-more in Barrett-surveillance": Care Evaluation of Barrett's Patients With Low-Risk in Whom Endoscopic Surveillance is Stopped. The BLISS Project
Brief Title: "Less-is-more in Barrett-surveillance" Care Evaluation of Barrett's Patients With Low-Risk in Whom Endoscopic Surveillance is Stopped. The BLISS Project.
Acronym: BLISS
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Nederlandse Barrett REgistratie Stichting (Unknown)
Responsible Party: Principal Investigator, Sanne van Munster, Doctor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: BLISS01
Record Dates: First submitted 2025-01-26; First posted 2025-01-31 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Barrett Esophagus; Barrett Esophagus Adenocarcinoma
Keywords: Barrett Esophagus; Esophageal cancer; Appropriate care; Endoscopic surveillance
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Discontinued endoscopic surveillance — Endoscopic surveillance is discontinued for eligible patients in line with the new guideline revision, and patients are then followed in this prospective cohort

SUMMARY:
Rationale:

Until recently, the conventional strategy outlined by both national and international guidelines for managing non-dysplastic (ND) Barrett esophagus (BE), involved endoscopic surveillance at 3 to 5 year intervals, aiming to reduce mortality from esophageal adenocarcinoma (EAC) through early detection and treatment. However, scientific evidence that supports the benefits in EAC-specific and/or overall survival, or that shows cost-effectiveness, is lacking. This has led to a re-evaluation of surveillance practices, particularly for NDBE patients at low risk of progression to EAC. For this reason, and in light of the 'NVMDL knowledge agenda,' a recent adjustment has been made to the Dutch guideline, recommending discontinuation of endoscopic surveillance for low-risk NDBE patients, hypothesizing that discontinuing endoscopic surveillance in low-risk NDBE patients will not lead to a relevant increase in the incidence of clinically significant EAC. This study aims to evaluate long-term outcomes of this guideline change.

Objective:

The primary objective is to evaluate the incidence of clinically apparent EAC after discontinuation of endoscopic surveillance in low-risk NDBE patients.

Study design: This is a nationwide, prospective, single-arm observational study with a minimum duration of 10 years. All patients in the Netherlands, eligible for study participation, will be approached and, upon signing informed consent, included in this care evaluation project. Baseline information will be collected from endoscopy and pathology reports and the electronic patient files. During follow-up, data will be collected from existing registries, including the national pathology database named Pathologisch-Anatomisch Landelijk Geautomatiseerd Archief (PALGA), the national statistics database named: Central Bureau van Statistiek (CBS), Integraal Kankercentrum Nederland (IKNL), and if necessary, additional information will be collected from electronic patient files in patient's hospital or the general practitioner.

On an annual basis, study outcomes will be evaluated and reviewed by a DSMB according to pre-defined stopping rules.

Study population:

All low-risk NDBE patients in the Netherlands in whom endoscopic surveillance will no longer be indicated based on the new Dutch guideline recommendations will be included. This includes patients with (1) BE with a maximum extent <5cm in length; (2) without (a history of) dysplasia; and (3) without a family history for EAC. A family history of EAC is defined as at least one first-degree relative with esophageal cancer.

Main study parameters/endpoints:

Primary study endpoint: the annual incidence of patients with clinically apparent EAC during a minimum follow-up of 10 years. Clinically apparent EAC is defined as one of the following:

* EAC related death, and/or
* EAC that exceeds boundaries for curative endoscopic treatment, defined as any symptomatic EAC that undergoes (1) palliative treatment; (2) esophagectomy; (3) chemotherapy; (4) radiotherapy; (5) immunotherapy; and/or (6) non-endoscopic therapy otherwise.

Two separate cohorts will be identified; (1) patients with an endoscopic surveillance history at the moment of study inclusion; and (2) patients with newly diagnosed NDBE at the moment of study inclusion. The primary endpoint will be evaluated separately in both cohorts. The power calculation will be based on the primary endpoint evaluation only in cohort 2, since cohort 1 is prone to selection bias.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

This registry that evaluates outcomes of regular clinical care, imposes minimal burden on participants. Subjects are not exposed to procedures or interventions. Data collection is based on existing national databases and medical records. Participants will provide informed consent for inclusion in the database, to ensure that patients understand the study's scope and their rights, with no further obligations for active involvement. Of note, discontinuation of endoscopic surveillance is standard practice according to the guideline. The current studies passively evaluates the outcomes, and patients only provide informed consent for inclusion in the registry. If a patient does not sign the informed consent form, the patient is not included in the registry, still, endoscopic surveillance for this patient will be discontinued.

Also robust measures will be implemented to ensure strict adherence to data protection regulations and safeguard participants' privacy and confidentiality. The primary focus remains on upholding ethical standards and minimizing any potential risks to participants while still be able to monitor relevant outcomes

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to be included in this study, a subject must meet all of the following criteria:

* Histological diagnosis of non-dysplastic Barrett's esophagus (NDBE).
* Barrett's esophagus segment with a maximum length of less than 5 cm (Prague classification M<5).
* At least one adequate, high-quality upper endoscopy with assessment of the Barrett segment performed according to existing guidelines, as evaluated by the referring endoscopist. A high-quality endoscopy is defined as: adequate imaging with high-resolutoin endoscope with sampling performed according to the Seattle protocol, and in absence of LA grade C or D reflux esophagitis. The endoscopist determines whether the last endoscopy was of high-quality. If this was not the case, the endoscopist may decide to schedule a new encoscopy.
* No recent history of confirmed indefinite for dysplasia (IND) or confirmed LGD, defined as no LGD and/or IND in the last 2 years and not in the last endoscopy.No history of HGD or cancer in BE
* Age ≥55 years and ≤75 years at the moment of inclusion.
* Informed consent provided by the patient or legal guardian.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* BE with (history of) dysplasia, either:

  * Prior cancer
  * Prior HGD
  * Confirmed LGD or IND in the last 2 years or during the last endoscopy
* Patients with an endoscopically visible lesion
* Patients with active reflux esophagitis LA grade C or D
* Patients with Barrett's esophagus with a maximum extent <1cm in length with currently already no surveillance indication.
* Patients with a family history of esophageal adenocarcinoma, defined as at least one first-degree relative with adenocarcinoma of the esophagus or gastric cardia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with low-risk Barrett esophagus
Sampling Method: Non-Probability Sample
Enrollment: 3156 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2038-02-07 (Estimated); Study Completion 2038-02-07 (Estimated)

PRIMARY OUTCOMES:
Clinical esophageal adenocarcinoma | 10 years
  Number of patietns with EAC related death, and/or EAC exceeding boundaries for endoscopic treatment EAC that exceeds boundaries for curative endoscopic treatment, defined as any symptomatic EAC that undergoes (1) palliative treatment; (2) esophagectomy; (3) chemotherapy; (4) radiotherapy; (5) immunotherapy; and/or (6) non-endoscopic therapy otherwise.

CONTACTS AND LOCATIONS:
Locations (1):
- Antoni van Leeuwenhoek - Centrum voor Vroegdiagnostiek (Barrett Coordination Centre), Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided